CLINICAL TRIAL: NCT01978990
Title: Assessment of a Health Informatics System on Insulin-treated Diabetic Patients
Status: Withdrawn | Type: Observational
Why Stopped: financial issues
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0406-13- HMO-CTIL
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2017-03

CONDITIONS: Type 1 or 2 Diabetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetes Management System , blood glucose

SUMMARY:
Modern medicine provides many solutions that are intended to help control the patient's blood glucose level: insulin and other medications to lower it, glucose tablets or glucagone to raise it when it gets dangerously low, glucometers to quickly measure the blood glucose level, pumps and pens to inject insulin or other injectable medicine, etc.The objective of this trial is proving the concept and the feasibility of using a medical informatics system comprised of computer hardware, software and a smartphone application to achieve better outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or 2 diabetics diagnosed at least 12 months prior to study enrollment.
2. Treated with insulin (basal only or basal + bolus) for at least 6 months prior to study enroment.
3. HbA1c lower than 12% With or without other anti-diabetic drugs.
4. 18-80 years of age.
5. Male or female.
6. Own an Android phone.
7. Able to handle mobile applications, technology-friendly
8. Able and willing to understand and comply with the study procedures.
9. Provide signed written and informed consent form prior to enrolment in the study.

Exclusion Criteria:

1. Using an insulin pump.
2. Pregnant or planning to be pregnant within the period of the study.
3. Active substance abuse.
4. Psychosis or schizophrenia under active care.
5. Uncorrected severe hearing or visual impairment.
6. Any other condition that is not acceptable to the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 or 2 diabetics diagnosed at least 12 months prior to study enrollment
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Recommendation accuracy | three months
  Recommendation accuracy: over 80% correspondence between the corrective actions recommended by the system and the corrective actions decided upon by the physician.